CLINICAL TRIAL: NCT03715114
Title: A Double-blind, Randomized, Placebo Controlled Single and Multiple Dose Study to Assess the Safety and Pharmacokinetics of Sodium Oligo-mannurarate (GV-971) Capsule in Healthy Chinese Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Oral Sodium Oligo-mannurarate (GV-971) in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRC-C1826
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Pharmacokinetics; Safety
MeSH Terms: interventions — GV-971

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GV-971 900 mg (Experimental): 900 mg oral
  Interventions: Drug: GV-971
- GV-971 1200 mg (Experimental): 1200 mg oral
  Interventions: Drug: GV-971
- GV-971 1500 mg (Experimental): 1500 mg oral
  Interventions: Drug: GV-971
- Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GV-971 — Oral GV-971
  Other Names: Sodium Oligo-mannurarate
  Arms: GV-971 1200 mg; GV-971 1500 mg; GV-971 900 mg
Drug: Placebo — Oral Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and pharmacokinetics of GV-971 capsules after oral a single or multiple doses of 900 mg, 1200 mg and 1500 mg in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects;
2. Age：≥18 and ≤40 on the date signing informed consent;
3. Body mass index (BMI): 19-26 kg/m2 and the weight ≥50 kg for male and ≥45 kg for female；
4. Subjects are able to understand the study procedures and methods, and willing to strictly comply with the protocol and give written informed consent.

Exclusion Criteria:

1. Subjects may be allergic to GV-971 in the opinion of the investigator;
2. With diseases which could impact on the absorption, distribution, metabolism and excretion (ADME) of study drugs or protocol adherence in the opinion of the investigator (such medical disorder/disease may relate to cardiovascular, liver, kidney, digestive, immune, blood, endocrine, metabolic, cancer, neuropsychiatric,etc );
3. Blood donation of ≥400 mL or severe blood lose and the volume of blood loss ≥400 mL within 12 weeks prior to screening;
4. Participation in any investigational drug or medical instrument study within 3 months prior to screening;
5. Use of any prescription medicine or herbal remedy, over the counter medication or dietary supplements such as vitamin, calcium within 2 weeks prior to screening;
6. Smoking more than 10 cigarettes a day, drugs or alcohol abuse within 6 months prior to screening;
7. Use of heparin, alginic sodium diester , mannose ester within 4 weeks prior to screening；
8. Clinically significant abnormalities in physical examination and laboratory test results or 12-lead ECG, etc. in screening;
9. Clinically significant abnormalities in Chest X-ray or abdominal B-ultrasound examination;
10. Positive seurology screen for Hepatitis B( HBsAg), Hepatitis C(HCV), HIV and USR unheated serum reagin test;
11. Vegetarian or person with dietary restrictions;
12. Subjects able to father a child are unwilling to use highly effective physical form of birth control from the trial period until 3 months after the completion of study;
13. Any other reasons that the subject is not eligible for participation in the study in the opinion of the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 2 day and 7 day
  Cmax will be determined after oral 900 mg, 1200 mg and 1500 mg of GV-971
Half life time (T1/2) | 2 day and 7 day
  T1/2 will be determined after oral 900 mg, 1200 mg and 1500 mg of GV-971
Area under the plasma concentration versus time curve (AUC) | 2 day and 7 day
  AUC will be determined after oral 900 mg, 1200 mg and 1500 mg of GV-971
Time to the peak drug concentration (Tmax) | 2 day and 7 day
  Tmax will be determined after oral 900 mg, 1200 mg and 1500 mg of GV-971

SECONDARY OUTCOMES:
Adverse Event (AE) | 7 days
  AE occurred after oral 900 mg, 1200 mg and 1500 mg of GV-971

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, MD, Principal Investigator — Shanghai Xuhui Center hospital
Locations (1):
- Phase-I Clinical Research Unit at Shanghai Xuhui Center hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No